CLINICAL TRIAL: NCT01042925
Title: A Phase 1/2 Study of XL147 (SAR245408) Administered in Combination With Trastuzumab or Paclitaxel and Trastuzumab in Subjects With Metastatic Breast Cancer Who Have Progressed on a Previous Trastuzumab-Based Regimen
Brief Title: Study of XL147 (SAR245408) in Combination With Trastuzumab or Paclitaxel and Trastuzumab in Subjects With Metastatic Breast Cancer Who Have Progressed on a Previous Trastuzumab-based Regimen
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARD11439; XL147-203 (Other: (other study code))
Record Dates: First submitted 2010-01-04; First posted 2010-01-06 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: HER2 positive breast cancer; breast cancer; breast tumors; human mammary carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — XL147; Trastuzumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): XL147 in combination with trastuzumab
  Interventions: Drug: XL147 (SAR245408); Biological: trastuzumab
- Arm 2 (Experimental): XL147 in combination with trastuzumab and paclitaxel
  Interventions: Drug: XL147 (SAR245408); Biological: trastuzumab; Drug: paclitaxel

INTERVENTIONS:
Drug: XL147 (SAR245408) — administered orally once daily as tablet(s)
Biological: trastuzumab — administered by IV once every 3 weeks
  Other Names: Herceptin
Drug: paclitaxel — administered by IV once every week
  Arms: Arm 2

SUMMARY:
Phase 1 of this study will evaluate the maximum tolerated dose (MTD) of XL147 when given in combination with trastuzumab (Herceptin) and in combination with trastuzumab and paclitaxel. After the MTD is established for each combination (Phase 2), subjects will be enrolled to evaluate the preliminary efficacy and safety of these combinations in metastatic HER2 positive breast cancer. Both trastuzumab and paclitaxel are used in the treatment of metastatic breast cancer (MBC), but patients can develop resistance.

The link between PI3K mutations and trastuzumab resistance has been seen in breast cancer patients. This suggests that inhibitors of the PI3K/PTEN pathway may have the potential to restore sensitivity to trastuzumab. Similarly, introduction of activated mutant forms of PI3K has been shown to transform and confer paclitaxel resistance to immortalized breast epithelial cells. XL147 is a potent and selective inhibitor of PI3K and inhibits phosphorylation of multiple downstream components of PI3K/PTEN signaling. Therefore, XL147 may have utility in the treatment of trastuzumab resistant/refractory and HER2-positive MBC when administered in combination with trastuzumab alone or with trastuzumab and paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* The subject has pathologically and radiologically confirmed metastatic HER2 positive breast cancer (Stage IV disease). Subjects must have received and progressed on at least one prior trastuzumab-containing regimen for metastatic disease. For subjects in Arm 2, they must also have received at least one prior taxane-containing regimen.
* The subject has at least one lesion that is not within a previously radiated field and measurable on computerized tomography (CT) or magnetic resonance imaging scan (MRI)
* The subjects enrolled in Phase 2 must be willing to undergo a biopsy of the primary tumor or a tumor metastasis at baseline, if tumor tissue is amenable to biopsy
* The subject's primary tumor and/or metastatic lesion must overexpress HER2
* For subjects enrolled in Phase 2: samples from archival or fresh tissue, or a tissue block of the subject's tumor.
* The subject has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* The subject has adequate organ and marrow function
* The subject is capable of understanding the informed consent and complying with the protocol and has signed the informed consent document prior to any study-specific screening procedures or evaluations being performed.
* Sexually active subjects must agree to use a medically-accepted barrier method of contraception during the course of the study and for 3 months following discontinuation of study treatments. For subjects using oral contraceptives, a barrier method must be used in addition to the oral contraceptive
* Subjects of childbearing potential must have a negative pregnancy test at screening and enrollment

Exclusion Criteria:

* The subject has previously been treated with a selective inhibitor of PI3K and / or AKT
* Certain restrictions on prior therapies apply
* The subject has not recovered from toxicity due to prior therapy to Grade ≤ 1 or to pre-therapy baseline
* The subject has untreated, symptomatic, or progressive brain metastases. Any corticosteroid use for brain metastases must have been discontinued without the subsequent appearance of symptoms for ≥4 weeks prior to first study treatment
* The subject has prothrombin time/International Normalized Ratio (PT/INR) or partial thromboplastin time (PTT) test results at screening that are ≥ 1.3 times above the laboratory upper limit of normal
* The subject has a diagnosis of uncontrolled diabetes mellitus
* The subject has uncontrolled significant intercurrent illness
* The subject has uncontrolled hypertension or other clinically significant cardiovascular disease
* The subject has left ventricular ejection fraction (LVEF) ≤ 50%
* The subject has a baseline corrected QT interval ≥ 460 ms
* The subject is currently receiving anticoagulation with therapeutic doses of warfarin (low-dose warfarin ≤ 1mg/day is permitted)
* The subject is pregnant or breastfeeding
* The subject is known to be positive for the human immunodeficiency virus (HIV) (a test for HIV at screening is not required)
* The subject has any other diagnosis of malignancy or evidence of malignancy (except non-melanoma skin cancer, in situ carcinoma of the cervix) within 2 years prior to screening for this study
* The subject has a previously identified allergy or hypersensitivity or is intolerant to components of any of the study treatment formulations
* The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of XL147 in combination with trastuzumab and in combination with trastuzumab and paclitaxel | safety assessments at weekly study visits
In Phase 1, the maximum tolerated dose (MTD) of XL147 when administered in combination with trastuzumab and in combination with trastuzumab and paclitaxel | assessed by weekly study visits
In Phase 2, objective tumor response | every 6 weeks

SECONDARY OUTCOMES:
Duration of response and progression-free survival (Phase 2) | every 6 weeks
Pharmacokinetics and pharmacodynamics of XL147 and trastuzumab when given in combination, and of XL147, trastuzumab, and paclitaxel when given in combination | assessed weekly, then every 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (9):
- United States (8):
  - Investigational Site Number 1537, Los Angeles, California
  - Investigational Site Number 1238, Fort Meyers, Florida
  - Investigational Site Number 1138, Boston, Massachusetts
  - Investigational Site Number 1330, Detroit, Michigan
  - Investigational Site Number 1150, New York, New York
  - Investigational Site Number 1151, The Bronx, New York
  - Investigational Site Number 1214, Nashville, Tennessee
  - Investigational Site Number 1246, Nashville, Tennessee
- Investigational Site Number 3413, Madrid, Spain